CLINICAL TRIAL: NCT06692829
Title: Investigation of the Effects of Robot-Assisted Therapy Added to Conventional Therapy on Hand Functions, Spasticity and Quality of Life in Patients With Chronic Stroke: A Randomized Controlled Trial
Brief Title: Robot-Assisted Therapy in Chronic Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAROBOT2
Record Dates: First submitted 2024-09-03; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Hemiplegia
Keywords: stroke; hemiplegia; robotic rehabilitation; hand function
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (Active Comparator): It was planned for the conventional therapy group to receive an exercise program consisting of 45 minutes of active, passive range of motion exercises and strengthening exercises, accompanied by a physiotherapist with at least 5 years of experience in stroke rehabilitation. A total of 20 treatment sessions will be applied 2 days a week.
  Interventions: Procedure: conventional rehabilitation
- Robot Assisted Therapy (Experimental): In addition to conventional therapy, the robotic therapy group was planned to receive robotic rehabilitation with a hand-finger robot [Amadeo (Tyromotion, Graz, Austria)] for 45 minutes, accompanied by a physiotherapist trained in robotic rehabilitation and with at least 5 years of experience. A total of 20 treatment sessions will be applied 2 days a week.
  Interventions: Procedure: robotic rehabilitation; Procedure: conventional rehabilitation

INTERVENTIONS:
Procedure: robotic rehabilitation — In addition to conventional therapy, the robotic therapy group was planned to receive robotic rehabilitation with a hand-finger robot [Amadeo (Tyromotion, Graz, Austria)] for 45 minutes, accompanied by a physiotherapist trained in robotic rehabilitation and with at least 5 years of experience. A total of 20 treatment sessions will be applied 2 days a week.
  Arms: Robot Assisted Therapy
Procedure: conventional rehabilitation — It was planned for the conventional therapy group to receive an exercise program consisting of 45 minutes of active, passive range of motion exercises and strengthening exercises, accompanied by a physiotherapist with at least 5 years of experience in stroke rehabilitation. A total of 20 treatment sessions will be applied 2 days a week.

SUMMARY:
Considering the paucity of studies on robotic hand therapy, larger-scale and long-term follow-up studies are needed. The aim in this study is to demonstrate the effectiveness of robot-assisted hand therapy in patients with chronic stroke and to compare this effectiveness in patients with different Brunnstrom stages.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of disability worldwide. Although mortality is decreasing, the number of people living with the effects of stroke has increased due to the increasing and aging population. It has been observed that 26% of patients have decreased basic daily living activities and 50% have decreased mobility after stroke.

Effective therapy in stroke rehabilitation should include repetitive, functional and task-specific exercises performed with high intensity and duration. In this context, in addition to traditional treatments, many new treatment approaches have come to the fore in recent years. Robot-assisted treatment (RAT) is one of these new treatment approaches. The use of robotic technology in rehabilitation has gained importance especially in the last 15 years and developments in this regard continue to increase. RAT is an innovative approach that includes intensive, repeatable, interactive and personalized applications.

This technology-based treatment increases the efficiency of rehabilitation care with its features of intensity, interaction, flexibility and adaptability to the patient performance and needs. It has no significant side effects and is well tolerated by patients. In the literature on robot-assisted treatment, different robotic devices have been used in various studies and different treatment protocols have been applied. This treatment has been reported to provide significantly greater improvement in function compared to conventional usual care. Studies in the literature on RAT demonstrate the feasibility of using these technologies in large patient groups.

The most common and devastating consequence of post-stroke disability is functional disability in the upper extremity. The functional prognosis of the lower extremity is generally better than the upper extremity after stroke. 20-30% of patients can walk normally, and 75% can reach some stage of ambulation. However, only 5% of patients return to normal upper extremity function, while 23-43% show inadequate functional recovery. Therefore, upper extremity rehabilitation requires more time and effort than lower extremity rehabilitation.

Bertani et al. In their published meta-analysis, they stated that robot-assisted rehabilitation is more effective in improving upper extremity motor function, especially in patients with chronic stroke, compared to conventional therapy. Amadeo (Tyromotion, Graz, Austria), an end-effector robotic rehabilitation device designed for hand rehabilitation, has shown feasibility and preliminary efficacy for stroke in the subacute phase. A randomized controlled trial with 17 patients compared conventional occupational therapy with Amadeo robotic therapy and after forty sessions, both groups showed significant improvement, but robotic intervention caused a greater improvement in hand function as measured by Fugl-Meyer and Motricity Index. Robotic hand therapy has started to take its place in routine rehabilitation protocols today. Considering the scarcity of studies on robotic hand therapy, it has been seen that larger-scale and long-term follow-up studies are needed. The aim in this study is to demonstrate the effectiveness of robot-assisted hand therapy in patients with chronic stroke and to compare this effectiveness in patients with different Brunnstrom stages.

ELIGIBILITY:
Inclusion Criteria:

* who were 3 months post-CVA
* whose health status was suitable for rehabilitation
* who could understand commands with a mini mental test score of 15 and above.

Exclusion Criteria:

* Patients with persistent upper extremity pain on the hemiplegic side (VAS>40)
* severe spasticity in the hand (MAS≥3)
* contracture in the hand
* fracture or surgery on the hemiplegic side within the last 6 months
* botulinum toxin injection into the upper extremity within the last 6 months
* skin ulcers
* brainstem or cerebellar lesions
* neglect or apraxia
* severe visual defects
* severe depression

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Brunnstrom Staging | Before treatment (T0) At the end of the treatment (10. week) (T1)
  is a test that evaluates the motor development of hemiplegic patients. In this test, the neurophysiological recovery process of the hemiplegic patient is defined as 6 stages. According to this staging, the lowest stage is stage 1 (flaccid, no voluntary movement stage), and the highest stage is stage 6 (isolated joint movement stage). In the Brunnstrom staging, the hand, upper extremity and lower extremity are evaluated separately.
Modified Ashworth Scale | Before treatment (T0) At the end of the treatment (10. week) (T1)
  Spasticity was planned to be evaluated with the Modified Ashworth Scale (MAS). In MAS, patients are evaluated over 5 points. 0 indicates no increase in muscle tone, and 4 indicates that the extremity is rigid in the flexion and extension directions.
Fugl Meyer Upper Extremity Assessment Questionnaire | Before treatment (T0) At the end of the treatment (10. week) (T1)
  The Fugl-Meyer Upper Extremity Motor Assessment Scale (FMUE Scale) was developed to quantitatively assess sensorimotor recovery after stroke. It was prepared based on Brunnstrom's stages of motor recovery. The FMUE Scale consists of 33 items, each scored from 0 to 2, where 0 = cannot perform, 1 = partially performs, and 2 = fully performs. The total score is 66.
ABILHAND Stroke Hand Function Questionnaire | Before treatment (T0) At the end of the treatment (10. week) (T1)
  ABILHAND Hand Questionnaire was developed in 1998 to measure the hand skill perceived by the patient. It contains 23 questions about how much difficulty the patient has in performing the activities. One of the options impossible (0 points), difficult (1 point), easy (2 points) is marked. The total score is 46.

SECONDARY OUTCOMES:
Mini Mental Test | Before treatment (T0) At the end of the treatment (10. week) (T1)
  The Mini Mental State Examination is a widely used cognitive screening test. The total score is 30 points. It has been stated that scores below 15 indicate low cognitive function, scores between 15-26 indicate moderate, and scores above 26 indicate high cognitive level. Turkish validity studies have been conducted in the normal population and in patients with traumatic brain injury.
Stroke Impact Survey | Before treatment (T0) At the end of the treatment (10. week) (T1)
  The Stroke Impact Scale (SIS) is a stroke-specific health status measure. It consists of 59 items and 8 sections. The patient is asked to rate the difficulty experienced in completing each item in the past week on a five-point Likert scale. A score of one indicates that the patient was unable to complete the item, and a score of five indicates that the patient had no difficulty in completing it. It also includes a visual analog scale (0: No improvement, 100: Full improvement) regarding the perception of general recovery after stroke. Validity and reliability studies have been conducted in Turkish.
Stroke Specific Quality of Life Scale (SSQOL) | Before treatment (T0) At the end of the treatment (10. week) (T1)
  SSQOL is a stroke-specific, patient-centered quality of life measure. SSQOL contains 49 items and consists of 12 domains; mobility, energy, upper extremity function, work/production, mood, self-care, social roles, family roles, vision, language, thinking, and personality. Each domain consists of at least 3 items, and each item is evaluated on a 5-point Likert scale considering the past week. Higher scores reflect better function. It has been shown to be valid and reliable for the Turkish population.